CLINICAL TRIAL: NCT01385605
Title: Analysis of Toxins in Follicle Fluid From Women With Unfulfilled Pregnancy
Brief Title: Analysis of Toxins in Follicle Fluid
Status: Completed | Type: Observational
Sponsor: Infertility Treatment Center Dortmund (Other)
Collaborators: TU Dortmund University (Unknown); Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Toxins FF 2015
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Environmental Exposure to Harmful Algae and Toxins; Female Subfertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — follicular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- female patients: ICSI treatment because of male subfertility

SUMMARY:
Environmental pollutants might be jointly responsible for increase of infertility among women. Especially endocrin active substances seem to be of particular importance. These substances are chemicals which interfere with the physiological system of humans and animals. They have a negative impact on the endocrine system and disturb the functions of organs whose hormones regulate the male and female reproductive system.

It is known that exposition to these chemicals lead to subfertility, infertility, raised abortions, birth defects and ovarian malfunction.

Additionally it was shown that human embryos have a decreased cleavage rate after IVF when developing from oocytes with elevated concentrations of environmental pollutants.

In this study the main focus concentrates on Nonylphenols (NP). Follicular fluids of women with subfertility will be analyzed by a newly developed principle including HPLC and NMR-Spectroscopy. This enables quantitative and qualitative analysis of enantiomers of NP.

The results will allow risk estimations for several endocrine active substances, especially NP.

Additionally conclusions concerning the correlation between thes substances and subfertility can be drawn.

DETAILED DESCRIPTION:
Exposure to environmental toxins may be responsible for female infertility. In particular substances known as endocrine disrupting chemicals (EDCs) may play a crucial role. These environmental toxins are either synthetic chemicals used in industry, agriculture or pharmacy, or natural chemicals found in food. Thus, exposure to EDCs can occur at different ways, e.g. drinking of contaminated water, breathing of contaminated air, or simple food intake. Despite most EDCs exhibit a long half-life, continuous accumulation of endocrine active substances will occur globally. In addition, low water-solubility and extremely high lipid-solubility promoted the accumulation within the human organism.

Consequently, EDCs may harm human health. It is known that EDCs lead to the disruption of the physiological system and that endocrine active substances interfere with the endocrine homeostasis. Moreover, EDCs alter organs that regulate male and female hormonal regulation crucial for reproduction fitness. Sterility and infertility, dysfunctional ovaries and an increased risk of abortions are discussed as critical consequences of EDC exposure.

It was shown that some endocrine active substances are present in the follicle fluid of women with unfilled pregnancy. Oocytes from follicles with an increased concentration of environmental toxins exhibit a reduced developmental potential. Additionally, women with an increased level of the EDC Bisphenol A tend to exhibit an increased risk of aborts.

Nonylphenol (NP) belongs to the class of endocrine active substances and are of special importance due to their high longevity and toxic characteristics. Nonylphenol is a multi-compound mixture that becomes generated as a by-product after degeneration of nonylphenol-ethoxylates (NPE) due to biological wastewater treatment. NPE are components of several cleaning agents, emulsifiers, dispersing agents and pesticides. NP is a mixture that consists mainly of para-substituted mono-alkylphenols with different isomeric nonyl-groups. Despite their high persistence and toxicity, exposure to NP induces alterations of the endocrine homeostasis in water organism, bird and mammals. NP can potentially bind to different hormone receptors (e.g. estrogen receptors, progesteron receptors and androgen receptors) and induce or modulate hormone-dependent downstream pathways. The influence regarding the reproductive fitness is much higher in females compared to males.

In the planned study, the follicle fluid will be analyzed in particular for the appearance of NP. Analysis will be done at the Institute of environmental research (Dortmund) in the group of Prof. Spiteller. Basis of this analysis is a chiral gas chromatography - mass spectroscopy that is optimized for the qualitative and quantitative assessment of NP isomers. For further details, see trial design and research setting.

Until now, two preliminary test series were done with at all 34 test persons. Within the first series of measurement, four patients exhibited an increased NP concentration in the follicle fluid (13.7 to 20.9 ng/g compared to 2.1 to 9 ng/g). In the second test series, the NP concentration was less prominent in all analyzed patients (average about 1 ng/ml), but detection of NP was still possible. Thus, NP was detected in all of the analyzed follicle fluid samples. However, the different NP concentration among all tested patients claims certainly the question, whether and how different concentration induce biological effects. The analysis of a large proband cohort regarding the appearance of NP within the follicle fluid facilitates the possibility to estimate a risk appraisal in patients with an unfilled pregnancy. Several parameters will be included for the evaluation: number of MII oocytes, fertilization rate, embryo quality, pregnancy rate, implantation rate and rate of abortions. Despite the duration of infertility and the number of previous IVF cycles will be considered, it is feasible to determine a correlation between the appearance of NP within the follicle fluid and the unfilled desire to have children.

ELIGIBILITY:
Inclusion Criteria:

* healthy females without sterility factors

Exclusion Criteria:

* job-related exposition to pollutants
* low responder

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female patients seeking ICSI treatment because of male subfertiliy
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2015-08; Primary Completion 2020-06-30 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 14 days after ICSI treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Dieterle, Principal Investigator — Infertility Treatment Center Dortmund
Locations (1):
- Infertility treatment center Dortmund, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bullach A, Trapphoff T, Zuhlke S, Spiteller M, Dieterle S. Impact of Nonylphenols and Polyhalogenated Compounds in Follicular Fluid on the Outcome of Intracytoplasmic Sperm Injection. Reprod Sci. 2021 Aug;28(8):2118-2128. doi: 10.1007/s43032-021-00472-y. Epub 2021 Feb 23. PMID 33620705